CLINICAL TRIAL: NCT07025551
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of MK-8527 in Participants With Mild and Moderate Hepatic Impairment
Brief Title: A Clinical Study of MK-8527 in Participants With Mild and Moderate Hepatic Impairment (MK-8527-015)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 8527-015; MK-8527-015 (Other: MSD)
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Impairment; Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mild Hepatic Impairment (Group 1) (Experimental): All participants will receive a single dose of MK-8527 on Day 1.
  Interventions: Drug: MK-8527
- Moderate Hepatic Impairment (Group 2) (Experimental): All participants will receive a single dose of MK-8527 on Day 1.
  Interventions: Drug: MK-8527
- Healthy (Group 3) (Experimental): All participants will receive a single dose of MK-8527 on Day 1.
  Interventions: Drug: MK-8527

INTERVENTIONS:
Drug: MK-8527 — Oral administration

SUMMARY:
The purpose of this study is to learn what happens to MK-8527 in a person's body over time (a pharmacokinetic [PK] study). Researchers will compare what happens to MK-8527 in the body when it is given to healthy participants and participants with mild and moderate hepatic (liver) impairment.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

All participants:

* Is a continuous non-smoker or moderate smoker (≤ 10 cigarettes per day or equivalent) for at least 3 months prior to dosing
* Has body mass index (BMI) ≥ 18.0 and ≤ 40.0 kg/m^2

Participants with Mild HI (Group 1) and Moderate HI (Group 2):

* Has mild or moderate hepatic impairment
* Has a diagnosis of chronic, stable, hepatic insufficiency with features of cirrhosis due to any etiology
* Is generally in good health with the exception of HI

Healthy Control Participants (Group 3):

- Healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, and ECGs

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

All participants:

* Has a history of cancer (malignancy)
* Has positive results for human immunodeficiency virus (HIV)
* Has had major surgery and/or donated or lost significant volume of blood within 56 days prior to dosing

Participants with Mild HI (Group 1) and Moderate HI (Group 2):

* With the exception of HI, has a history or presence of clinically significant medical or psychiatric condition or disease
* Is positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb)
* Is positive for Hepatitis C Virus (HCV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration versus time curve from 0 to the time of the last quantifiable sample (AUC0-last) of MK-8527 | Predose and at designated timepoints up to 168 hours post dose
  Plasma samples will be collected at pre-specified timepoints to determine the AUC0-last of MK-8527.
Area under the concentration versus time curve from 0 to infinity (AUC0-inf) of MK-8527 | Predose and at designated timepoints up to 168 hours post dose
  Plasma samples will be collected at pre-specified timepoints to determine the AUC0-inf of MK-8527.
Maximum Observed Concentration (Cmax) of MK-8527 | Predose and at designated timepoints up to 168 hours post dose
  Plasma samples will be collected at pre-specified timepoints to determine the Cmax of MK-8527.
Time to Maximum Concentration (Tmax) of MK-8527 | Predose and at designated timepoints up to 168 hours post dose
  Plasma samples will be collected at pre-specified timepoints to determine the Tmax of MK-8527.
Apparent Terminal Half-life (t1/2) of MK-8527 | Predose and at designated timepoints up to 168 hours post dose
  Plasma samples will be collected at pre-specified timepoints to determine the t1/2 of MK-8527.
Apparent Clearance (CL/F) of MK-8527 | Predose and at designated timepoints up to 168 hours post dose
  Plasma samples will be collected at pre-specified timepoints to determine the CL/F of MK-8527.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-8527 | Predose and at designated timepoints up to 168 hours post dose
  Plasma samples will be collected at pre-specified timepoints to determine the Vz/F of MK-8527.

SECONDARY OUTCOMES:
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 29 days
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 29 days
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
AUC0-inf of MK-8527-triphosphate (TP) in peripheral blood mononuclear cell (PBMCs) | Predose and at designated timepoints up to 672 hours post dose
  Blood samples will be collected to determine the AUC0-inf of MK-8527-TP.
Area under the concentration versus time curve from 0 to 672 hours after dosing (AUC0-672hrs) of MK-8527-TP in PBMCs | At designated timepoints pre dose and up to approximately 672 hours post dose
  Blood samples will be collected to determine the AUC0-672 of MK-8527-TP.
Cmax of MK-8527-TP in PBMCs | Predose and at designated timepoints up to 672 hours post dose
  Blood samples will be collected to determine the Cmax of MK-8527-TP.
Concentration at 672 Hours (C672) of MK-8527-TP in PBMCs | Predose and at designated timepoints up to 672 hours post dose
  Blood samples will be collected to determine the C672 of MK-8527-TP.
Tmax of MK-8527-TP in PBMCs | Predose and at designated timepoints up to 672 hours post dose
  Blood samples will be collected to determine the Tmax of MK-8527-TP.
T1/2 of MK-8527-TP in PBMCs | Predose and at designated timepoints up to 672 hours post dose
  Blood samples will be collected to determine the Tmax of MK-8527-TP.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Arizona Clinical Trials ( Site 0001), Chandler, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com